CLINICAL TRIAL: NCT00809497
Title: A Randomized, Multi-centre, Double-blind and Placebo Controlled Clinical Study of the Propionyl-L-carnitine Hydrochloride Tablets
Brief Title: A Clinical Study on Efficacy & Safety Profile of Propionyl-L-carnitine Tablets for Peripheral Arterial Diseases
Acronym: PLC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Collaborators: Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PLC-LZ00108; SFDA-2006L03870
Record Dates: First submitted 2008-12-16; First posted 2008-12-17 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2008-03

CONDITIONS: Peripheral Arterial Disease
Keywords: PLC for treatment of peripheral arterial diseases
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Propionyl-L-carnitine Tablets — 500mg tablets, oral administration of 2g daily
  Other Names: DROMOS, ST261

SUMMARY:
The main objective of this study is to evaluate the effectiveness and safety of the propionyl-L-carnitine hydrochloride tablets among Chinese population in comparison with the placebo, for treatment of the peripheral arterial diseases (intermittent claudication) with oral supplementation of 2g daily for a 4 months continuous administration.

DETAILED DESCRIPTION:
This is a randomized, multi-centre, double-blind and placebo controlled clinical study. Propionyl-L-Carnitine (PLC) is a kind of natural derivative of L-Carnitine (LC) and is produced in the body and concentrated by 90% in the skeletal muscle and myocardium via an enzyme-mediated reaction involving propionyl-CoA and LC. For oral adminsitration, PLC shows that the decrease of the leg muscle carnitine of the PAD patient appears to correlate with poor exercise performance. It has recently been shown that the severity of the impairment in walking distance is correlated with the impairment in carntine metabolism at the muscle level. 2g daily of PLC supplementation can significantly improve the walking ability in patients with IC with a maximum walking capacity between 50 and 250 meters on the treadmill.

ELIGIBILITY:
Inclusion Criteria:

* The variability between the two standardized claudication tests during the wash-out period must be <20%, as assessed by the formular: (Highest MWD-Lowest MWD)/(Lowest MWDxx100%)
* At the last visit during the wash-out period, the ABI at rest must be ,0.9

Exclusion Criteria:

* with rest pain, ulceration, and/or gangrene
* PAD of a non-atherosclerotic nature
* Aortic or lower extremity arterial surgery, angioplasty, or lumbar sympathectomy within 6 months; any above ankle level amputation. Any type of major surgery during the last three months.
* Except PAD, any concomitant disease that can limit patients' performance in the treadmill exercise.
* with angina (at rest or activity) or any symptom which is sufficiently severe to discontinue the treadmill exercises.
* Myocardial infarction within 6 months
* Severe cerebral dysfunction
* Type I diabetes (Stable type II diabetes can also be included)
* alcohol or drug abused history within 3 months
* Medium or severe anaemia (Hb,90g/L)
* Platelets <100 x 10 9/L
* Bleeding diathesis
* Renal insufficiency or hepatic function laboratory test result>1.5 normal value
* Treatment with LC or carnitien derivatives in the past 3 months
* Pregnancy, lactation, fertility without adequate protest against pregnancy
* Reject to sign the informed consent form

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 239 (Actual)
Dates: Start 2008-05; Primary Completion 2009-09 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To compare the difference between pre-and post-the treatment of each group | 4 months

SECONDARY OUTCOMES:
Statistically describe the variance of ABI, CT and other indexes at the end of 4th month | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jianxin Li, MD, Principal Investigator — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital Capital Medical University, Beijing, Beijing Municipality, China